CLINICAL TRIAL: NCT01294436
Title: A Long Term Open Label Study to Evaluate the Safety and Efficacy of Dapagliflozin as Monotherapy or Combination Therapies With Anti-diabetic Drugs in Japanese Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Evaluate Safety as Mono or Combination Therapies With Anti-diabetes Mellitus Drugs in Japanese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1692C00012
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-11

CONDITIONS: Type2 Diabetes; High Blood Sugar
Keywords: Phase3; Clinical trial; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus, Type 2 | interventions — dapagliflozin

ARMS (1):
- Open label treatment (Experimental)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Oral Dose 5 or 10 mg

SUMMARY:
This is a long term, single arm, open label study to evaluate the safety and efficacy of dapagliflozin as monotherapy or in combination therapy with other anti diabetic drug in Japanese subjects with type 2 diabetes mellitus who have inadequate blood sugar control on diet and exercise or on other anti-diabetic treatment will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Men or women age ≥20 years old (Either gender needs to be 40% or higher of total number of treated subjects)
* diagnosed with type2 DM ; ≥6.5% and ≤10% at 1 week before treatment started

Exclusion Criteria:

* Type 1 diabetes mellitus,
* FPG >240 mg/dL before treatment started
* Subjects who have history of unstable or rapidly progressing renal disease
* Subjects who have severe hepatic insufficiency and/or significant abnormal liver function
* Significant cardiovascular history

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jisin Yang, MD, Study Director — AstraZeneca KK
Locations (38):
- Japan (38):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Owariasahi, Aichi-ken
  - Research Site, Toyohashi, Aichi-ken
  - Research Site, Hirosaki, Aomori
  - Research Site, Niihama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Itoshima, Fukuoka
  - Research Site, Yukuhashi, Fukuoka
  - Research Site, Annaka, Gunma
  - Research Site, Ōta, Gunma
  - Research Site, Aki-gun, Hiroshima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sanuki, Kagawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kamakura, Kanagawa
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Zushi, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Sendai, Miyagi
  - Research Site, Matsumoto, Nagano
  - Research Site, Osaka, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Ōtsu, Shiga
  - Research Site, Atami, Shizuoka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Komatsushimachō, Tokushima
  - Research Site, Chiyoda City, Tokyo
  - Research Site, Chūō, Tokyo
  - Research Site, Mitaka, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Shibuya City, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Taitō City, Tokyo
  - Research Site, Takaoka, Toyama
  - Research Site, Toyama, Toyama
  - Research Site, Ube, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 28-Feb-2011; Last subject last visit: 15-Sep-2012; 1030 participants were enrolled in 56 Japanese centers. 728 Japanese men and women aged >=20 years with inadequate glycemic control (HbA1c levels of 6.5% to 10.0% prior to study treatment) with diet and exercise were treated.
Pre-assignment Details: A 6-week wash-out period was applicable only for subjects with ongoing anti-diabetic treatment at enrolment. A 4-week lead-in period was applicable for all subjects.
Groups:
- Monotherapy: Dapagliflozin 5/10 mg only
- All Combination Therapies: Dapagliflozin 5/10 mg in combination with any anti-diabetic drugs
Period: Overall Study
Arm/Group | Monotherapy | All Combination Therapies
Started | 249 | 479
Completed | 221 | 409
Not Completed | 28 | 70
Not completed — Adverse Event | 10 | 17
Not completed — Withdrawal by Subject | 11 | 28
Not completed — subject no longer meets study criteria | 5 | 20
Not completed — poor/non-compliance | 2 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all subjects who received at least one dose of study medication and who provided any safety records.
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy | All Combination Therapies | Total
Number analyzed (Participants) | 249 | 479 | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.40) | 57.2 (10.06) | 57.5 (10.18)
Age, Customized [Number; unit: participants]
  < 65 years | 182 | 365 | 547
  65 - <75 years | 55 | 102 | 157
  >= 75 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 211 | 314
  Male | 146 | 268 | 414
Region of Enrollment [Number; unit: participants]
  Japan | 249 | 479 | 728
Body Weight [Mean (Standard Deviation); unit: kg] | 67.77 (13.437) | 67.40 (14.529) | 67.52 (14.157)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.72 (4.196) | 25.61 (4.440) | 25.64 (4.355)
Seated Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 127.5 (13.73) | 125.8 (14.13) | 126.4 (14.01)
HbA1c [Mean (Standard Deviation); unit: Percent] | 7.53 (0.761) | 7.82 (0.865) | 7.72 (0.842)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 140.29 (25.355) | 147.35 (29.097) | 144.93 (28.057)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Adverse Events
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to adverse events
Time Frame: Long-term treatment up to 52 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 249 | 479
Percentage of participants | 79.1 | 72.4

2. Primary Outcome: Proportion of Participants With Serious Adverse Events
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to serious adverse events
Time Frame: Long-term treatment up to 52 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 249 | 479
Percentage of participants | 5.6 | 3.1

3. Primary Outcome: Proportion of Participants With At Least One Episode of Hypoglycemia
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to occurrence of hypoglycemia
Time Frame: Long-term treatment up to 52 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 249 | 479
Percentage of participants | 2.4 | 4.0

4. Primary Outcome: Mean Change in Hematocrit
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in hematocrit
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
Percent | 2.17 (0.1396) | 2.00 (0.1115)

5. Primary Outcome: Mean Change in Alanine Aminotransferase (ALT)
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in alanine aminotransferase
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
U/L | -7.1 (0.955) | -5.4 (0.622)

6. Primary Outcome: Mean Change in Aspartate Aminotransferase (AST)
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in aspartate aminotransferase
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 405
U/L | -3.9 (0.695) | -2.6 (0.410)

7. Primary Outcome: Mean Change in Blood Urea Nitrogen (BUN)
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in blood urea nitrogen
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
mg/dL | 2.4 (0.250) | 2.3 (0.168)

8. Primary Outcome: Mean Change in Magnesium
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in magnesium (1 mEq/L equivalent to 0.50 mmol/L)
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
mEq/L | 0.05 (0.0074) | 0.05 (0.0064)

9. Primary Outcome: Mean Change in Serum Uric Acid
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in serum uric acid
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
mg/dL | -0.61 (0.0578) | -0.50 (0.0374)

10. Primary Outcome: Mean Change in Seated Heart Rate
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in pulse
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
beats per minute (bpm) | -0.4 (7.52) | 0.2 (7.95)

11. Primary Outcome: Mean Change in Seated Diastolic Blood Pressure
Description: To evaluate the safety and tolerability of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in blood pressure
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
mmHg | -2.9 (8.16) | -2.1 (8.73)

12. Primary Outcome: Mean Change in Seated Systolic Blood Pressure
Description: as for outcome 11
Time Frame: Baseline to Week 52
Population: Safety Analysis Set, participants with non-missing baseline and week 52 values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 220 | 407
mmHg | -5.2 (11.68) | -3.9 (13.03)

13. Other Pre Specified Outcome: Mean Change in HbA1c Levels
Description: To evaluate the efficacy of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in HbA1c
Time Frame: Baseline to Week 52
Population: Full Analysis Set, participants with non-missing baseline and week 52 (LOCF) value
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 249 | 477
Percent | -0.66 (11.68) [-0.75 to -0.57] | -0.68 (13.03) [-0.75 to -0.62]

14. Other Pre Specified Outcome: Mean Change in Body Weight
Description: To evaluate the efficacy of long-term treatment up to 52 weeks with the dosing regimen of dapagliflozin, where it started with 5 mg and titrated up to 10 mg depending on participant's condition of glycemic control, in regard to the change in body weight
Time Frame: Baseline to Week 52
Population: Full Analysis Set, participants with non-missing baseline and week 52 (LOCF) value
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Monotherapy | All Combination Therapies
Number analyzed (Participants) | 249 | 477
kg | -2.58 (11.68) [-2.87 to -2.30] | -2.06 (13.03) [-2.31 to -1.81]

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 52-week open-label treatment period plus 4/30 days or up to follow-up visit if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Monotherapy | All Combination Therapies
Serious Adverse Events (participants affected / at risk) | 14/249 | 15/479
Other Adverse Events (participants affected / at risk) | 71/249 | 126/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=249) | All Combination Therapies (N=479)
AGE RELATED MACULAR DEGENERATION (Eye disorders) | 1 | 0
CATARACT (Eye disorders) | 1 | 1
RETINAL DETACHMENT (Eye disorders) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLONIC POLYP (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
CHRONIC SINUSITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 3
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
TACHYCARDIA PAROXYSMAL (Cardiac disorders) | 0 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=249) | All Combination Therapies (N=479)
NASOPHARYNGITIS (Infections and infestations) | 63 | 116
POLLAKIURIA (Renal and urinary disorders) | 13 | 13

LIMITATIONS AND CAVEATS:
In the efficacy analysis, for participants who did not complete 52-week treatment period LOCF (last observation carried forward) was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.